CLINICAL TRIAL: NCT07173738
Title: An Open Label, Three Period, Fixed Sequence Study to Assess the Pharmacokinetics, Safety and Tolerability of Concurrent Doses of BIA 5-1058 and Furosemide in Healthy Subjects Under Fasting Conditions.
Brief Title: Pharmacokinetics, Safety and Tolerability of Concurrent Doses of BIA 5-1058 and Furosemide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BIA-51058-111; 2017-002807-93 (EudraCT Number)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension (PAH); BIA 5-1058; Zamicastat; Furosemide; Dopamine ß-hydroxylase (DßH) inhibitor; BIAL
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BIA 5-1058 (Experimental): Period 1: Single oral dose of BIA 5-1058 400 mg
  Interventions: Drug: BIA 5-1058
- Furosemide (Experimental): Period 2: 40 mg furosemide (single oral dose)
  Interventions: Drug: Furosemide
- BIA 5-1058 and Furosemide (Experimental): Period 3: 40 mg furosemide (single oral dose) concomitant with a single oral dose of BIA 5-1058 400 mg
  Interventions: Drug: BIA 5-1058 and Furosemide

INTERVENTIONS:
Drug: BIA 5-1058 — During treatment period 1, a single oral dose of BIA 5-1058 (400 mg) will be administered on the morning of day 1, following an overnight fast of at least 10 h.
  Other Names: Period 1
  Arms: BIA 5-1058
Drug: Furosemide — During treatment period 2, a single oral dose of furosemide (40 mg) will be administered on the morning of day 1, following an overnight fast of at least 10 h.
  Other Names: Period 2
  Arms: Furosemide
Drug: BIA 5-1058 and Furosemide — During treatment period 3, a single oral dose of both investigational medicinal product (IMPs) BIA 5-1058 (400 mg) concomitantly with furosemide (40 mg) will be administered on the morning of day 1, following an overnight fast of at least 10 h.
  Other Names: Period 3
  Arms: BIA 5-1058 and Furosemide

SUMMARY:
The purpose of this study is:

* To assess the effect of BIA 5 1058 400 mg on furosemide pharmacokinetics (PK).
* To assess the effect of furosemide 40 mg on the PK of BIA 5 1058.

DETAILED DESCRIPTION:
This was an open-label, single-dose, fasted, 3-periods, fixed-sequence study separated by a washout period of 10 days or more in healthy volunteers.

Each healthy subject will participate in the study for approximately 3 months, including a 28-day screening period, 3 periods of 3.5 days and 4 nights (inpatient) with each dosage separated by a 10 day washout period and a follow-up visit. The inpatient period will be from Day -1 to Day 4 morning. Dosing will occur on Day 1 and subjects will remain in the clinic until 72 hours (h) after administration.

A Follow up visit will be performed 14 ± 2 days after discharge of the last period.

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated informed consent form before any study-specific screening procedure is performed;
2. Males and Females subjects aged 18 to 55 years, inclusive;
3. Non-smoker or ex-smokers for at least 3 months prior to screening;
4. Body mass index (BMI) between 18 and 30 kg/m2, inclusive;
5. Subject with no clinically significant history of previous allergy / sensitivity to BIA 5-1058/furosemide or any of the excipients contained within the IMP(s);
6. Negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus antibodies (HCV Ab) and anti-human immunodeficiency virus antibodies (HIV-1 and HIV-2 Ab) at screening;
7. Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period;
8. Healthy as determined by the Investigator based on medical history, physical examination, , vital signs (systolic blood pressure (SBP) ≥ 90 mmHg and ≤ 140 mmHg, diastolic blood pressure (DBP) ≥ 50 mmHg and ≤ 90 mmHg) and digital 12-lead electrocardiogram (ECG));
9. Clinical laboratory test results clinically acceptable at screening and admission to each treatment period;

   If male:
10. Male subjects and female partner willing to use 2 effective methods of contraception, i.e., established method of contraception + condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of IMP.
11. Refraining from donating sperm throughout the study and for 3 months after the last dose of IMP;

    If female:
12. No childbearing potential by reason of surgery or at least 1 year post-menopause (i.e., 12 months post last menstrual period), or menopause confirmed by follicle-stimulating hormone (FSH) testing;
13. If of childbearing potential, using an effective non-hormonal method of contraception [intrauterine device; condom or occlusive cap (diaphragm or cervical or vault caps) with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he is the sole partner of that subject] for all the duration of the study and for 3 months after the last dose of IMP;
14. Negative serum pregnancy test at screening and negative urine pregnancy test on admission of each treatment period).

Exclusion Criteria:

1. Any personal or family history of haemostatic disorder;
2. Consumption of more than 21 units (14 units for female subjects) of alcohol a week [1 unit corresponds to 1 glass of 12% wine (10 cl), 1 glass of 45% pastis (2.5 cl), 1 glass of 40% whisky (2.5 cl), 1 glass of 12% champagne (10 cl), 1 glass of 18% aperitif drink (7 cl) or one 25-cl glass of 5% beer];
3. Use of nicotine replacement products such as patches, gum and/or electronic cigarettes within 3 months prior to the screening visit;
4. Significant infection or known inflammatory process at screening or admission to each treatment period;
5. Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period;
6. Symptomatic orthostatic hypotension [drop of > 20 mmHg in SBP and/or > 10 mmHg] in DBP when moving from supine to standing position, together with other symptoms, e.g. dizziness
7. Previous use of BIA 5-1058;
8. Use of any investigational drug or participation in any clinical trial within 90 days or 5 half-life times, whichever is longer,
9. Participation in more than 4 clinical trials within the 12 months prior to screening;
10. Donation or reception of any blood or blood products within the 3 months prior to screening;
11. Vegetarians, vegans or other medical dietary restrictions;
12. Not able to communicate reliably with the Investigator;
13. Unlikely to co-operate with the requirements of the study;
14. Use of medicines within 28 days of initiation of treatment that may affect the safety or other study assessments, in the Investigator's opinion or intake of any of the prohibited medications.
15. Clinically relevant history or presence of respiratory, gastrointestinal, hepatic, renal, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders;
16. Clinically relevant surgical history that could interfere with the pharmacokinetics of the trial medications;
17. No medication will be permitted throughout the study, except for medications to treat adverse events (AEs).
18. Subject has an abnormal hepatic function based on an overall assessment by the Investigator regarding medical history, physical examination and laboratory tests of hepatic function (ALT > 1times the upper limit of normal (ULN), aspartate transaminase (AST) > 1times the ULN and total bilirubin > 1times the ULN [confirmed by subsequent repeat]), as judged by the Principal Investigator. If a laboratory assessment is outside of the reference range at the local laboratory at the Screening Visit or baseline, the assessment may be repeated once as soon as possible and in any cases before enrolment to rule out laboratory error.
19. Any clinically relevant findings in the laboratory tests, including any abnormality in the coagulation tests;
20. History of alcoholism or drug abuse;
21. Females who are currently breast feeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 3 months
  Will be calculated from the treatment periods 1, 2 and 3, days 1 to 4, BIA 5-1058 and furosemide concentration-time data
Time to Cmax (Tmax) | Up to 3 months
  Will be calculated from the treatment periods 1, 2 and 3, days 1 to 4, BIA 5-1058 and furosemide concentration-time data
Elimination rate constant (kel) | Up to 3 months
  Will be calculated from the treatment periods 1, 2 and 3, days 1 to 4, BIA 5-1058 and furosemide concentration-time data
Terminal elimination half-life (t1/2) | Up to 3 months
  Will be calculated from the treatment periods 1, 2 and 3, days 1 to 4, BIA 5-1058 and furosemide concentration-time data
Area under the concentration-time curve (AUC) from time of dosing to last measurable concentration (AUC0-t) | Up to 3 months
  Will be calculated from the treatment periods 1, 2 and 3, days 1 to 4, BIA 5-1058 and furosemide concentration-time data
AUC extrapolated to infinity (AUC0-inf) | Up to 3 months
  Will be calculated from the treatment periods 1, 2 and 3, days 1 to 4, BIA 5-1058 and furosemide concentration-time data
Clearance (CL/F) | Up to 3 months
  Will be calculated from the treatment periods 1, 2 and 3, days 1 to 4, BIA 5-1058 and furosemide concentration-time data
Volume of distribution (Vz/F) | Up to 3 months
  Will be calculated from the treatment periods 1, 2 and 3, days 1 to 4, BIA 5-1058 and furosemide concentration-time data
AUC% extrapolated (residual area) | Up to 3 months
  Will be calculated from the treatment periods 1, 2 and 3, days 1 to 4, BIA 5-1058 and furosemide concentration-time data

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, Dr, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd (Simbec), Merthyr Tydfil, United Kingdom